CLINICAL TRIAL: NCT06713616
Title: Comparative Effectiveness of Racemic Ketamine Versus Esketamine (Spravato®) for Depression
Brief Title: PCORI Comparative Effectiveness Study-Esketamine (Spravato) vs. Ketamine-Equivalence Study
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Samuel Wilkinson, Associate Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000037121; 23-005287 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2024-11-27; First posted 2024-12-03 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2024-11

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Esketamine

STUDY DESIGN:
Intervention Model Description: This study is a randomized phase 3 drug treatment study. Subjects will be randomized, in randomly varying blocks of no more than 8 at each site, to receive either esketamine (Spravato®) or intravenous ketamine. This study is unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Racemic Ketamine (Experimental): Ketamine will be given intravenously. Per FDA guidance, the max dose of ketamine will be 60mg per day, with a total lifetime limit of 8 doses. Ketamine will be infused over 40 minutes.
  Interventions: Drug: Racemic ketamine
- Spravato (Esketamine) (Experimental): Spravato® (Esketamine) will be given intranasally. For esketamine, the dose will be between 56 and 84mg, according to the FDA label for the drug. Allowances will be made for patients who have difficulty tolerating these doses to be dosed at 28mg in subsequent treatment sessions.
  Interventions: Drug: Spravato (Esketamine)

INTERVENTIONS:
Drug: Racemic ketamine — Ketamine will be given intravenously. Per FDA guidance, the max dose of ketamine will be 60mg per day, with a total lifetime limit of 8 doses. Ketamine will be infused over 40 minutes.
  Arms: Racemic Ketamine
Drug: Spravato (Esketamine) — Spravato® (Esketamine) will be given intranasally. For esketamine, the dose will be between 56 and 84mg, according to the FDA label for the drug. Allowances will be made for patients who have difficulty tolerating these doses to be dosed at 28mg in subsequent treatment sessions.
  Arms: Spravato (Esketamine)

SUMMARY:
The purpose of this study is to compare the relative effectiveness, acceptability, and side effects of ketamine delivered through an IV (a drip into the arm) which is not currently FDA approved for use in the treatment of treatment-resistant depression (TRD) and Esketamine (Spravato®), taken as a nasal spray which has received FDA approval for use in the treatment of treatment-resistant depression (TRD) in the treatment of patients with treatment-resistant depression (TRD). The study will look at the following:

* How well the treatment helps with symptoms of depression (effectiveness),
* How comfortable and willing people are to use the treatment (acceptability), and
* How well people can deal with any side effects from the treatment (tolerability).

The study will also examine factors that may predict which treatment works better for certain patients.

DETAILED DESCRIPTION:
This non-inferiority, multi-site, comparative effectiveness study will utilize a randomized design. Individuals with treatment resistant depression (TRD) will be randomized (1:1) to Spravato® or IV ketamine. This 5-year multisite comparative effectiveness study will enroll 400 total patients (~200 per group).

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Adults ages 18 or older
* Diagnosis of major depressive disorder that is refractory to two or more antidepressant trials
* Moderate or severe depression based on an initial MADRS score ≥ 25
* Judged appropriate for ketamine or esketamine by clinician, independent of potential study participation
* A female participant must be:

  a. Not of childbearing potential*, OR b. Of childbearing potential and practicing a highly effective method of contraception (failure rate of <1% per year when used consistently and correctly) and agrees to remain on a highly effective method while receiving study intervention and until 1 week after last dose - the end of relevant systemic exposure. The investigator will evaluate the potential for contraceptive method failure (e.g., noncompliance, recently initiated) in relationship to the first dose of drug. Acceptable methods of contraception are: i. combined (estrogen and progestogen containing) hormonal or progestogen-only hormonal contraception associated with inhibition of ovulation (oral, transdermal, or intravaginal) ii. intrauterine device (IUD) iii. intrauterine hormone-releasing system (IUS) iv. bilateral tubal occlusion/ligation v. male partner with a bilateral vasectomy with documented aspermia or a bilateral orchiectomy vi. male or female condom with spermicide, diaphragm, or sponge with spermicide (Note: Use of condom as the sole method of contraception is not considered to be a highly effective method of contraception).
* A female participant must agree not to donate eggs (ova, oocytes) or freeze for future use for the purposes of assisted reproduction during the study * We will consider women to be of childbearing potential if they are within 2 years of menopause (within 3 years since last menstrual period) and have not had a hysterectomy, bilateral oophorectomy, or other definitive surgical intervention.

Exclusion Criteria:

* Diagnosis of bipolar disorder or psychotic disorder (i.e., schizophrenia, schizoaffective disorder)
* Other psychiatric comorbidities are permitted so long as depression is the predominant diagnosis
* Active or recent (within 12 months) substance use disorder (other than nicotine)
* Pregnant or lactating women
* Intracerebral hemorrhage or aneurysmal vascular disease
* Hypersensitivity to ketamine, esketamine or any of the excipients
* Known family history of ketamine use disorder
* Prior known ketamine use disorder as well as subjects for whom study participations will result in more than 8 lifetime exposures to ketamine (e.g., prior exposure to ketamine, prior recreational use with ketamine)
* Uncontrolled hypertension, as demonstrated by a blood pressure of greater than 145 / 90 at screening visit. (Pre-treatment blood pressure will be permitted to be 150 / 95 to allow for "whitecoat" hypertension on treatment visits 1-8.)
* Known cardiovascular and cerebrovascular conditions that are associated with an increased risk related to ketamine or esketamine administration (including space-occupying CNS lesions). This includes those prospective participants who undergo EKG and are shown to have an abnormality that would put them at increased risk related to treatment.
* Known condition for which an acute rise in blood pressure would pose a serious risk.
* Arteriovenous malformation
* Positive urine toxicology at screening visit, except for substances that are prescribed (i.e., benzodiazepines, stimulants). Given the extended length of time between exposure and negative toxicology screen, a positive screen for THC will not be exclusionary unless the pattern of use and clinical evaluation are indicative of cannabis use disorder. Cannabis used within 24 hours of dosing is exclusionary.
* Positive alcohol breathalyzer at screening or clinical signs of intoxication
* The patient is unable to arrange for someone to drive them home after each treatment session; patients who are unwilling to refrain from driving and operating machinery on treatment days until the next day following sleep will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Self-Reported Effectiveness | 30 days
  defined as the change in depression severity after 8 treatments, as assessed by the 16-item, patient-reported outcome, Quick Inventory of Depression Symptomatology (QIDS-SR16), at the end of one-month of treatment. Scale ranges from 0 - 27 with higher scores indicating worse depression.

SECONDARY OUTCOMES:
Clinician-Reported Effectiveness | baseline until end of treatment (4 weeks)
  change in Montgomery-Asberg Depression Rating Scale (MADRS) score. Scale ranges from 0-60 with higher scores indicating worse depression.
Response | baseline until end of treatment (4 weeks)
  defined as a ≥50% decrease from baseline to end of week 4 on the Quick Inventory of Depression Symptomatology (QIDS-SR16). The proportion and number of participants with response will be compared between groups.
Remission | baseline until end of treatment (4 weeks)
  defined as a total score of ≤ 5 on the Quick Inventory of Depression Symptomatology (QIDS-SR16). The proportion and number of participants with remission will be compared between groups.
Suicidal Ideation and Behavior | baseline until end of treatment (4 weeks)
  The Columbia-Suicide Severity Scale Rating (C-SSRS) will be collected to examine any comparative differences in suicidal ideation. Scale ranges from 0-5 (for suicidal ideation) with higher scores indicating worse ideation. Scale for behavior measures counts of suicide behaviors.
Level of Disability | baseline until end of treatment (4 weeks)
  The Sheehan Disability Scale (SDS) will be used to assess any changes in patient disability levels associated with the treatments. The SDS is a patient rated discretized analog measure of functional disability in work, social and family life. Score for each subscale ranges from 0-10, with higher scores indicating worse disability.
Quality of Life | baseline until end of treatment (4 weeks)
  defined as changes in quality of life, as assessed by the Quality of Life in Depression Scale (QLDS). The QLDS will assess changes in the quality-of-life factors in relation to antidepressant treatments. The score ranges from 0-34, with higher scores indicating worse quality of life.
Utilization of Healthcare Resources | end of treatment (4 weeks)
  Measure using the Health Resource Utilization Questionnaire to track all cause healthcare utilization by assessing patients visits to all forms of healthcare providers and settings and tracking the use of other health related resources. In specific, group comparisons on specific types of patient visits (e.g., therapy visits, hospitalizations, ED visits) will be made. The scale measures counts of healthcare visits.
Acceptability | end of treatment (4 weeks after baseline)
  The 9-item Treatment Satisfaction Questionnaire for Medication (TSQM-9) will be used as the key secondary outcome measure. The TSQM-9 is a validated tool for assessing patient satisfaction with treatment and covers the domains of effectiveness, convenience, and global satisfaction. Each domain is scored from 0-100 with lower scores indicating lower satisfaction. Behavioral measures will be used to assess treatment acceptability by comparing dropout rates and missed visits between the two treatment options.
Patient and Clinician Global Severity and Improvement | baseline until end of treatment (4 weeks)
  Global improvement of depression will be assessed with the Clinician and Patient Global Impression-Severity/Improvement indices. These are simple measures for clinicians and patients to provide information on overall depression severity and improvement with treatment. The scale ranges from 1-7 with higher scores indicating worse depression.
Tolerability and Safety | baseline until end of treatment (4 weeks)
  Tolerability will be based on group comparison of number of patients who experience adverse events of special interest. These include vomiting, dysphoric reactions, and clinically meaningful elevations in blood pressure and/or heart rate during the treatment session.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Wilkinson, MD, Principal Investigator — Samuel.Wilkinson@yale.edu
Locations (6):
- United States (6):
  - Mood Institute, Milford, Connecticut
  - Yale School of Medicine, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - University of Michigan, Ann Arbor, Michigan
  - LifeStance Health, Moore, Oklahoma
  - Houston Center for Advanced Psychiatric Treatment, Bellaire, Texas

IPD SHARING:
Plan to Share IPD: No